CLINICAL TRIAL: NCT06284018
Title: Effect of Progressive Muscle Relaxation Exercises Versus Pilates Exercises on Postnatal Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Ahmed Safy Eldeen Mahmoud, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: postnatal low back pain
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Low Back Pain
Keywords: Progressive muscle relaxation exercises; Pilate's exercises; Low back pain.; post natal period; relaxation exercises
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: intervention The design of the study was randomized controlled study. The patients were divided randomly into two equal groups (A&B). Group A consisted of thirty postnatal women. They were treated by progressive muscle relaxation exercises three times per week for 4 weeks. Group B consisted of thirty postnatal women. They were treated by pilates exercises three times per week for 4 weeks.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group1 (Experimental): Group A consisted of thirty postnatal women. They were treated by progressive muscle relaxation exercises three times per week for 4 weeks.
  Interventions: Other: Progressive Muscle Relaxation Exercises
- intervention group 2 (Experimental): Group B consisted of thirty postnatal women. They were treated by pilates exercises three times per week for 4 weeks.
  Interventions: Other: Pilates Exercises

INTERVENTIONS:
Other: Progressive Muscle Relaxation Exercises — * Focus on the targeted muscle group.
  * Take a slow, deep breath while squeezing on muscle group as hard as she can (not to the point of strain). Keep the muscle tensed for 5 seconds.
  Hands and arms, forehead ,Eyes and Cheek, Mouth and Jaw , Neck and Shoulder ,Stomach , Leg and Toes
  Arms: intervention group1
Other: Pilates Exercises — Pilates exercise program consisted of floor exercises on a rubber mat, including the following exercises: a- Pelvic Curl. b- Single-Leg Lift. c- Chest Lift. d- Supine Spine Twist. e- Basic Back Extension.
  Arms: intervention group 2

SUMMARY:
This study was conducted to compare between the effect of progressive muscle relaxation exercises and the effect of pilates exercises on postnatal low back pain

DETAILED DESCRIPTION:
Ethical approval was obtained from the Institutional Review Board of the Faculty of Physical Therapy, Cairo University, before starting this study [No: P.T.REC/012/003885]. The study's protocol was explained in detail to each woman who signed an informed consent form before starting this study. This work adhered to the principles outlined in the Declaration of Helsinki for the ethical conduct of research involving human subjects. It was carried out from June till September 2023

Sample Size Calculation:

Based on a pilot study, sample size was calculated according to the significant difference in the value of mean difference (pretreatments - post treatment values) of pain pressure algometer between progressive muscle relaxation exercises (2.01 ± 0.39) and pilates exercises (2.90 ± 0.24) groups in unpaired t test, with α=0.05, power of 80%, and an effect size of 0.74. So a sample size of 30 patients/per group would be required and increased to 35 women to allow for a 15% dropout rate (GPower 301 http:www.psycho.uni-duesseldorf.de) Randomization of sample selection was achieved using closed envelop way. Classification of the sample by simple random way into two groups equal in number, by using sixty closed envelop, each thirty envelop contained a name of a group from the two groups (Group A) or (Group B) and asking each woman to choose one envelop from them, each woman attended to the group according the name of the group written in her envelop. After randomization, they were divided into two groups equal in number

ELIGIBILITY:
Inclusion Criteria:

* ages were ranged from 25 to 35 years old and their body mass index (BMI) did not exceed 30kg/m2. They were postnatal by three months. The number of parity of all women was ranged from (1-3) times.

Exclusion Criteria:

* previous trauma to the spine, pelvis and lower limbs,
* previous history of spinal surgery (such as spinal fusion surgery, vertebroplasty, or - --kyphoplasty), congenital spinal deformities, history of spinal tumors, ankylosing spondylitis, osteoporosis other spondyloarthritis

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-24 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Pressure Algometer | period of treatment was 4 weeks
  Assessment of pressure pain thresholds is a valid and reliable clinical tool to evaluate the subjective perception of pain in response to application of pressure in low back pain patient. Pressure algometry is used in manual therapy to objectively quantify the pressure pain thresholds and it was shown that a predictable variation exists across various spinal levels from cervical to lumbar levels. The examiner determined the main 4 points of assessment (5 cm lateral to the spinous process of L3 and L5 bilaterally), the force of PA was gradually increased at a rate of 1 kg/s, by silently counting seconds while increasing pressure, then the patient was asked to tell the examiner when the pressure became painful while the examiner applied the pressure on the assessment points

SECONDARY OUTCOMES:
Oswestry Disability Index | period of treatment was 4 weeks
  ODI (P) is a reliable and valid instrument for measurement of disability related to low back pain in Punjabi population. It can be used both in research and clinical care settings in future Sandal, D., [12] . The 10 factors which constitute the ODI criteria for assessing patients' functional impairment are pain intensity, ease of personal care, lifting, working, sitting, standing, sleeping, sex life, social life and travelling. Each of the 10 questions was scored from 0 to 5, giving a maximum score of 50. The total score is then converted into a percentage by multiplying it by 2. Scores are stratified into severity:
  * 0-4: No disability
  * 5-14: Mild disability
  * 15-24: Moderate disability
  * 25-34: Severe disability
  * 35-50: Completely disabled

CONTACTS AND LOCATIONS:
Overall Officials: Hala M Emara, phd, Study Director — Cairo University
Locations (1):
- faculty of physical therapy: Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No